CLINICAL TRIAL: NCT04631185
Title: Antibiotics and Surgical Site Infection in Expander Based Breast Reconstruction Trial (ASSERT) A Multi-institutional Randomized Controlled Trial to Determine the Optimal Antibiotic Prophylaxis for Tissue Expander-based Breast Reconstruction
Brief Title: Surgical Site Infection and Antibiotic Use Study
Acronym: ASSERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Plastic Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSF 19-03-SSI Study
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Surgical Site Infection; Breast Reconstruction; Antibiotic Use
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPD (Arm A) (Active Comparator): Single pre-operative dose of intravenous antibiotics with intraoperative redosing (SPD): Intravenous cefazolin, a cephalosporin antibiotic, will be prescribed to all patients before surgery. All patients will receive one dose of antibiotic within 60 minutes prior to incision, and any intraoperative doses of antibiotics according to current recommendations based on the antibiotic's dosing and on operative time.
  Interventions: Drug: Single pre-operative dose of intravenous antibiotics with intraoperative redosing
- WPO (Arm B) (Experimental): The patients assigned to this arm will receive same pre-op and intraoperative antibiotics similar to SPD (Arm A). In addition, patients in this group will receive one week of post-operative antibiotics (WPO). The post-operative antibiotic will be a first generation Cephalosporin of their surgeon's choice.
  Interventions: Drug: Single pre-operative dose of intravenous antibiotics with intraoperative redosing; Drug: One week of post-operative antibiotics

INTERVENTIONS:
Drug: Single pre-operative dose of intravenous antibiotics with intraoperative redosing — Intravenous cefazolin, a cephalosporin antibiotic, will be prescribed to all patients before surgery. In case of allergy to cefazolin, intravenous clindamycin will be prescribed. For allergy to both antibiotics, an appropriate antibiotic should be chosen by the surgeon and documented. All patients will receive one dose of antibiotic within 60 minutes prior to incision, and any intraoperative doses of antibiotics according to current recommendations based on the antibiotic's dosing and on operative time.
Drug: One week of post-operative antibiotics — The patients will be prescribed one week of Cephalosporin Antibiotic (Keflex/Duricef/Other) of their surgeon's choice.
  Arms: WPO (Arm B)

SUMMARY:
This study is a prospective, multi-institutional, noninferiority, randomized control trial that will compare the efficacy of two antibiotic treatments in preventing SSI in patients receiving immediate breast reconstruction with tissue expanders (TE-BR). The patients will be randomly assigned to one of the two treatment groups. One group will receive a single dose of antibiotics just before surgery and if necessary, more doses during the surgery. The other group will receive the same treatment as the first group, along with an additional week of antibiotics after surgery. The study will assess the rates of SSI from the two groups. It will also assess the type, duration and method (oral vs. intravenous) of subsequent antibiotic use for patients who develop SSIs in each group.

DETAILED DESCRIPTION:
Among plastic surgeons, the clinical practice of prescribing postoperative prophylactic antibiotics following postmastectomy breast reconstruction with tissue expanders ranges widely from no postoperative antibiotics, to 5-7 days post-op, to antibiotics until the drains are removed. The Centers for Disease Control and Prevention (CDC) recommends a single preoperative antibiotic dose for clean and clean-contaminated procedures, even in the presence of a drain. With the CDC creating a national action plan to reduce unnecessary prophylactic antibiotics for clean non-contaminated cases by advocating use of only a single pre-operative dose of antibiotics (see: https://www.cdc.gov/drugresistance/pdf/national_action_plan_for_combating_antibotic-resistant_bacteria.pdf ) there is mounting pressure on the plastic surgery community to adopt this regimen of SSI prophylaxis. Because there are no definitive studies that provide sufficient or conclusive evidence to affect antibiotic practice patterns among plastic surgeons on a large-scale, plastic surgeons use a wide variety of protocols for their SSI prophylaxis, especially in implant-based breast reconstruction. Plastic surgeons have generally not adopted CDC guidelines because these recommendations were not based on studies in plastic surgery patients, and the use of foreign body implants underneath devitalized soft tissue can be associated with higher infection risks. Based on the literature and from self-reporting from ASPS membership, there is a wide range of prophylactic antibiotic use to prevent SSI from as little as one preoperative dose to many weeks of therapy; one week of post-operative antibiotics is the most common form. However, the Centers for Disease Control (CDC) recommends a single preoperative dose of antibiotics for clean cases, even in the presence of a drain. Prolonged antibiotic courses can lead to antibiotic complications and development of resistance.

Definitive studies to determine an optimal therapeutic strategy to prevent SSI in implant-based plastic surgical procedures are lacking. This study will address a dilemma in common plastic surgical operation: the use of post-operative antibiotics in prosthesis-based breast reconstruction.

The central hypothesis for this multi-institutional, prospective randomized control trial (RCT) is that a single pre-operative dose of intravenous antibiotics with intraoperative redosing (SPD) is no worse (noninferiority design) at preventing SSI in tissue expander-based breast reconstruction (TE-BR) than an additional week of post-operative antibiotic prophylaxis (WPO).

This trial will evaluate the efficacy of single preoperative dose versus one-week antibiotic regimens in preventing surgical site infection after tissue expander breast reconstruction. The investigators will assess the rates of SSI from the SPD vs. the WPO groups. They will assess the type, duration and method (oral vs. intravenous) of subsequent antibiotic use for patients who develop SSIs in each group. The study will also compare the readmission and premature expander removal rates due to SSI and the adverse antibiotic side effects in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older, undergoing unilateral or bilateral mastectomy (including breast cancer, any stage, or prophylactic) and immediate tissue expander reconstruction (including submuscular, submuscular and ADM, or pre-pectoral placement).

Exclusion Criteria:

* Breast cancer patients not undergoing mastectomy

  * Patients undergoing direct-to-implant reconstruction
  * Patients undergoing delayed reconstruction
  * Patients having autologous reconstruction
  * History of radiation to the breast or chest
  * History of previous breast reconstruction on the side of expander placement
  * Patients with serious existing systemic infection, defined as 2 or more of the following: Peripheral body temperature >38 degrees Celsius CRP >5g/L Leukocytes > 12,000/microliter at the time of enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Number of participants in each group who develop surgical site infection (SSI) within 30 days of index procedure. | Up to 30 days after the index procedure
  Surgical site infection as defined by CDC criteria within 30 days after the index procedure

SECONDARY OUTCOMES:
Number of participants in each group with antibiotic-related adverse events and the type of adverse events reported. | Up to 30 days after the index procedure
  Antibiotic-related adverse events, e.g. colitis, yeast infections, anaphylaxis, etc.
Number of participants in each group who develop an SSI or other complications after 30 days of index procedure. | Up to two years
  SSI beyond 30 days after the index procedure up to the time of tissue expander exchange (for an implant or flap)
Number of participants in each group who undergo premature tissue expander or implant removal. | From index procedure until expander removal
  Tissue expander or implant removal, per breast and per patient events will be calculated
Type, duration and route of antibiotic administration (Oral or Intravenous) in participants in each group who develop SSI/deep infections. | Up to two Years
  Antibiotic sensitivities in SSI/deep infections,
Comparison of any secondary infections, including resistant bacterial strains and yeast infections, in participants from the two groups who develop SSI. | Up to two Years
  Speciation of any cultures from wound or tissue samples derived from participants in each group who develop SSI will be performed
ER visit and hospital readmission rates among participants in both groups. | Up to two Years
  Length of hospitalization, need for surgery, extent of surgery (e.g. wound revision, loss of implant) will be assessed. ER visit and hospitalization rates will be recorded for comparison between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rohde, MD, MPH, Principal Investigator — Columbia University; Brian Gastman, MD, Principal Investigator — The Cleveland Clinic
Locations (5):
- United States (5):
  - The University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
The study sites will keep patient details under a study ID number, and not under the patient's name. Aggregate data shared between investigators will be coded and de-identified (except dates).